CLINICAL TRIAL: NCT05457231
Title: Effects of Specific Feedback Based on an In-depth Assessment Tool for Communication Skills Training Protocol in Occupational Therapy Interns
Brief Title: Effects of SF for CST Protocol in OT Interns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202001194B0
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Communication; Occupational Therapy
Keywords: communication skills; communication skills training; feedback; communication skills assessment; communication skills measure; occupational therapy; intern
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CST-SF group (Experimental): The feedback process was as follows. Feedback was given after each interview, including brief feedback and SF. Brief feedback was provided by the clinical instructor based on the Gap-Kalamazoo Communication Skills Assessment Form immediately after each interview. Within two weeks after the first and second interviews, the interns received SF from experts and clinical instructors based on the Communication Skills Measure for Therapist. The SF of the third interview could not be completed because the internship had ended.
  Interventions: Other: specific feedback based on an in-depth assessment tool for communication skills training

INTERVENTIONS:
Other: specific feedback based on an in-depth assessment tool for communication skills training — In addition to the specific feedback based on an in-depth assessment tool, four strategies modified from common strategies in the previous studies were incorporated into the intervention protocol, including lecture, patient interview, brief feedback, and self-reflection

SUMMARY:
Specific feedback is considered an important strategy in communication skills training (CST). However, the effects of specific feedback on communication skills have not been comprehensively investigated. Therefore, this study aimed to investigate the effects of specific feedback based on an in-depth assessment tool for CST (CST-SF) in occupational therapy interns' communication skills.

DETAILED DESCRIPTION:
A one-group pretest-posttest study was conducted. Thirty-six interns received CST-SF combined with patient interviews and brief feedback. Each intern completed three interviews with different patients. After the interviews, the interns were given brief feedback based on the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF) and specific feedback based on the Communication Skills Measure for Therapists. The first and last interviews were assessed by experts, clinical instructors, interns, and patients using the GKCSAF.

ELIGIBILITY:
Inclusion Criteria:

* fourth-year undergraduate students who had started their psychiatry internship

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Gap-Kalamazoo Communication Skills Assessment | Change from Baseline GKCSAF scores at 3 months
  The Gap-Kalamazoo Communication Skills Assessment (GKCSAF) is widely used in medical education to evaluate communication skills in patient interviews through observation and to provide immediate feedback

CONTACTS AND LOCATIONS:
Overall Officials: TZU-TING CHEN, Master, Principal Investigator — Chang Gung Memorial Hospital and Chang Gung University College of Medicine, Kaohsiung, Taiwan
Locations (1):
- Chang Gung Medical Hospital, Kaohsiung City, Niaosong Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillis AE, Morris MC, Ridgway PF. Communication skills assessment in the final postgraduate years to established practice: a systematic review. Postgrad Med J. 2015 Jan;91(1071):13-21. doi: 10.1136/postgradmedj-2014-132772. Epub 2014 Dec 2. PMID 25468984
- [Background] van Es JM, Schrijver CJ, Oberink RH, Visser MR. Two-dimensional structure of the MAAS-Global rating list for consultation skills of doctors. Med Teach. 2012;34(12):e794-9. doi: 10.3109/0142159X.2012.709652. Epub 2012 Sep 3. PMID 22938687
- [Background] Riess H, Kraft-Todd G. E.M.P.A.T.H.Y.: a tool to enhance nonverbal communication between clinicians and their patients. Acad Med. 2014 Aug;89(8):1108-12. doi: 10.1097/ACM.0000000000000287. PMID 24826853
- [Background] Epstein RM, Street RL Jr. Shared mind: communication, decision making, and autonomy in serious illness. Ann Fam Med. 2011 Sep-Oct;9(5):454-61. doi: 10.1370/afm.1301. PMID 21911765
- [Background] Fallowfield L, Jenkins V. Effective communication skills are the key to good cancer care. Eur J Cancer. 1999 Oct;35(11):1592-7. doi: 10.1016/s0959-8049(99)00212-9. PMID 10673967